CLINICAL TRIAL: NCT01207336
Title: Effect of Combined Anodal tDCS and Peripheral Nerve Stimulation on Motor Recovery in Acute Stroke
Brief Title: Combined tDCS+PNS After Acute Stroke
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C09-27; 2009-A01153-54 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischaemic Stroke
Keywords: stroke; rehabilitation; transcranial direct current stimulation; nerve stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: combined transcranial direct current stimulation and electrical peripheral nerve stimulation — tDCS: 1,2 mA 13 minutes rEPNS (radial nerve): 5 Hz, 0,7 x MT

SUMMARY:
Recent work showed that application of peripheral nerve and cortical stimulation independently can induce 10-15 % improvement in motor performance in patients with chronic stroke.

The purpose of this study was to compare in post-stroke hemiplegic patients the effect on motor recovery of one session of anodal transcranial direct current stimulation to the ipsilesional primary motor cortex (M1) combined with a peripheral radial nerve electrical stimulation (rEPNS) to the paretic hand repeated 5 successive days with the effect of the same peripheral nerve stimulation combined with sham tDCS.

Design: randomized, double-blind, parallel controlled clinical trial. Patients eligible for the study: Acute ischaemic stroke Primary outcome measure: Jebsen Taylor test Secondary outcome measures Nine peg hole test Hand tapping grip and wrist force Cortical excitability of Ipsilesional M1(TMS) Follow-up: 30 days

ELIGIBILITY:
Inclusion Criteria:

- first -ever ischemic stroke within 5-30 days a paresis of the arm/hand with NIHSS <15 age 35-85 years

Exclusion Criteria:

Pregnancy psychiatric disease patients with history of alcohol or drug abuse or severe depression patients with a severe language disturbances, particularly of receptive nature patients with increased intracranial pressure or serious cardiac disease patients with contraindication to TMS

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-08-30 (Actual); Study Completion 2012-08-30 (Actual)

PRIMARY OUTCOMES:
Jebsen Taylor test | 5-15-30 days

SECONDARY OUTCOMES:
Grip and wrist force Nine peg hole Cortical excitability ofIpsilesional M1 (TMS) | 5-15-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marion SIMONETTA-MOREAU, MDPhD, Study Director — Inserm; Imagerie cerebrale et handicaps neurologiques UMR 825; F-31059 Toulouse, France; François CHOLLET, MDPhD, Principal Investigator — Centre Hospitalier Universitaire de Toulouse; Pole Neurosciences; CHU Purpan, Place du Dr Baylac, F-31059 Toulouse Cedex 9, France
Locations (1):
- Centre d' Investigation Clinique de Toulouse et Hopitaux de Toulouse ( Purpan), Toulouse, France

REFERENCES:
- [Background] Loubinoux I, Dechaumont-Palacin S, Castel-Lacanal E, De Boissezon X, Marque P, Pariente J, Albucher JF, Berry I, Chollet F. Prognostic value of FMRI in recovery of hand function in subcortical stroke patients. Cereb Cortex. 2007 Dec;17(12):2980-7. doi: 10.1093/cercor/bhm023. Epub 2007 Mar 26. PMID 17389628
- [Background] Castel-Lacanal E, Gerdelat-Mas A, Marque P, Loubinoux I, Simonetta-Moreau M. Induction of cortical plastic changes in wrist muscles by paired associative stimulation in healthy subjects and post-stroke patients. Exp Brain Res. 2007 Jun;180(1):113-22. doi: 10.1007/s00221-006-0844-5. Epub 2007 Jan 31. PMID 17265041
- [Background] Castel-Lacanal E, Marque P, Tardy J, de Boissezon X, Guiraud V, Chollet F, Loubinoux I, Moreau MS. Induction of cortical plastic changes in wrist muscles by paired associative stimulation in the recovery phase of stroke patients. Neurorehabil Neural Repair. 2009 May;23(4):366-72. doi: 10.1177/1545968308322841. Epub 2008 Dec 5. PMID 19060132
- [Background] Conchou F, Loubinoux I, Castel-Lacanal E, Le Tinnier A, Gerdelat-Mas A, Faure-Marie N, Gros H, Thalamas C, Calvas F, Berry I, Chollet F, Simonetta Moreau M. Neural substrates of low-frequency repetitive transcranial magnetic stimulation during movement in healthy subjects and acute stroke patients. A PET study. Hum Brain Mapp. 2009 Aug;30(8):2542-57. doi: 10.1002/hbm.20690. PMID 19072894
- [Background] Celnik P, Paik NJ, Vandermeeren Y, Dimyan M, Cohen LG. Effects of combined peripheral nerve stimulation and brain polarization on performance of a motor sequence task after chronic stroke. Stroke. 2009 May;40(5):1764-71. doi: 10.1161/STROKEAHA.108.540500. Epub 2009 Mar 12. PMID 19286579
- [Background] Uy J, Ridding MC. Increased cortical excitability induced by transcranial DC and peripheral nerve stimulation. J Neurosci Methods. 2003 Aug 15;127(2):193-7. doi: 10.1016/s0165-0270(03)00142-0. PMID 12906948
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411